CLINICAL TRIAL: NCT05119855
Title: A Phase 3, Multicenter, Open-Label Study to Evaluate the Safety and Immunogenicity of 2-dose Regimens of 9vHPV and mRNA-1273 SARS-CoV-2 Vaccines Where the First Dose of Each Vaccine Are Given Concomitantly in Boys and Girls 9 to 11 Years of Age
Brief Title: Safety and Immunogenicity of 9-valent Human Papillomavirus (9vHPV) Vaccine Coadministered With Messenger Ribonucleic Acid (mRNA)-1273 Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) (COVID-19) Vaccine (V503-076)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-076; 2021-003591-13 (EudraCT Number)
Record Dates: First submitted 2021-11-10; First posted 2021-11-15 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Papillomavirus Infections; Coronavirus Disease (COVID-19)
MeSH Terms: conditions — Papillomavirus Infections; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; COVID-19 Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Concomitant Group (Experimental): Participants will receive Dose 1 of 9-valent human papillomavirus [Types 6, 11, 16, 18, 31, 33, 45, 52, 58] (9vHPV) vaccine administered into the left arm as an intramuscular (IM) injection, AND Dose 1 of the messenger ribonucleic acid (mRNA)-1273 vaccine administered into the right arm as an IM injection on Day 1; participants will then receive Dose 2 of the mRNA-1273 vaccine administered into the right arm as an IM injection at Month 1 and Dose 2 of the 9vHPV vaccine administered into the left arm as an IM injection at Month 6.
  Interventions: Biological: 9vHPV Vaccine; Biological: mRNA-1273 Vaccine
- Non-concomitant Group (Experimental): Participants will receive Dose 1 of the mRNA-1273 vaccine administered into the right arm as an IM injection on Day 1 and Dose 2 of the mRNA-1273 vaccine administered into the right arm as an IM injection at Month 1. Participants will then receive Dose 1 of the 9vHPV vaccine administered into the left arm as an IM injection at Month 2 and Dose 2 of the 9vHPV vaccine administered into the left arm as an IM injection at Month 8.
  Interventions: Biological: 9vHPV Vaccine; Biological: mRNA-1273 Vaccine

INTERVENTIONS:
Biological: 9vHPV Vaccine — 9-valent human papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) administered as a 0.5-mL intramuscular (IM) injection
  Other Names: V503; GARDASIL®9; SILGARD®9
Biological: mRNA-1273 Vaccine — mRNA-1273 50 mcg dose administered as a 0.25-mL IM injection
  Other Names: SARS-CoV-2 Vaccine; Moderna COVID-19 Vaccine

SUMMARY:
The purpose of this study to evaluate the safety and immunogenicity of a 2-dose regimen of 9vHPV vaccine, where the first dose is administered concomitantly with a first dose of a 2-dose regimen of mRNA-1273 vaccine versus nonconcomitant administration of 9vHPV and mRNA-1273 vaccines in boys and girls 9 to 11 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Has not yet had coitarche and does not plan on becoming sexually active during the vaccination period
* Participant or participant's legally acceptable representative can read, understand, and complete the electronic vaccination report card (eVRC).

Exclusion Criteria:

* Known allergy to any vaccine component
* History of severe allergic reaction that required medical intervention
* Thrombocytopenia or any coagulation disorder
* Has a history of myocarditis or pericarditis
* Has a history of a clinical or microbiological diagnosis of COVID-19 ≤90 days prior to Day 1 visit or history of multisystem inflammatory syndrome in children (MIS-C) at any time prior to Day 1 visit
* Females only: participant is pregnant
* Currently immunocompromised, or been diagnosed with immunodeficiency
* Had a splenectomy
* Receiving or has received immunosuppressive therapies within the last year
* Received any immunoglobulin product or blood-derived product within 3 months
* Received a marketed HPV vaccine or has participated in an HPV vaccine clinical trial

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (38):
- United States (38):
  - Cognitive Clinical Trials, LLC ( Site 0054), Phoenix, Arizona
  - Eclipse Clinical Research ( Site 0095), Tucson, Arizona
  - Children's Clinic of Jonesboro, PA ( Site 0044), Jonesboro, Arkansas
  - Preferred Research Partners Inc. ( Site 0092), Little Rock, Arkansas
  - Coast Clinical Research, LLC ( Site 0027), Bellflower, California
  - Ark Clinical Research ( Site 0098), Long Beach, California
  - Valley Clinical Trials Inc. ( Site 0004), Northridge, California
  - Medical Center for Clinical Research ( Site 0051), San Diego, California
  - Ark Clinical Research ( Site 0108), Tustin, California
  - Emerson Clinical Research Institute ( Site 0021), Washington D.C., District of Columbia
  - Accel Research Sites-DeLand Clinical Research Unit ( Site 0066), DeLand, Florida
  - Advanced Research for Health Improvement, LLC ( Site 0012), Immokalee, Florida
  - Acevedo Clinical Research Associates ( Site 0001), Miami, Florida
  - Alpha Science Research ( Site 0067), Miami, Florida
  - Advanced Research For Health Improvement LLC ( Site 0075), Naples, Florida
  - Comprehensive Clinical Research ( Site 0038), West Palm Beach, Florida
  - Atlanta Center for Medical Research ( Site 0055), Atlanta, Georgia
  - Mount Vernon Clinical Research ( Site 0053), Sandy Springs, Georgia
  - Clinical Research Prime ( Site 0088), Idaho Falls, Idaho
  - CBH Health ( Site 0019), Gaithersburg, Maryland
  - SKY Integrative Medical Center/SKYCRNG ( Site 0084), Ridgeland, Mississippi
  - Midwest Children's Health Research Institute ( Site 0003), Lincoln, Nebraska
  - Certified Research Associates ( Site 0090), Cortland, New York
  - Corning Center for Clinical Research ( Site 0091), Horseheads, New York
  - Carolina Institute for Clinical Research, LLC ( Site 0042), Fayetteville, North Carolina
  - M3 Wake Research, Inc. ( Site 0014), Raleigh, North Carolina
  - Dayton Clinical Research ( Site 0028), Dayton, Ohio
  - Thomas Jefferson University - Family and Community Medicine ( Site 0006), Philadelphia, Pennsylvania
  - WR-ClinSearch ( Site 0049), Chattanooga, Tennessee
  - DermResearch, Inc. ( Site 0056), Austin, Texas
  - South Texas Clinical Research ( Site 0024), Corpus Christi, Texas
  - South Texas Pediatric Research Group ( Site 0094), Del Rio, Texas
  - West Houston Clinical Research Services ( Site 0078), Houston, Texas
  - Next Level Urgent Care, LLC ( Site 0099), Houston, Texas
  - Milton Haber, M.D. ( Site 0069), Laredo, Texas
  - University of Texas Medical Branch ( Site 0026), League City, Texas
  - University of Utah ( Site 0076), Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City ( Site 0025), West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26855&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Concomitant Group: Participants received Dose 1 of 9-valent human papillomavirus [Types 6, 11, 16, 18, 31, 33, 45, 52, 58] (9vHPV) vaccine administered into the left arm as an intramuscular (IM) injection, AND Dose 1 of the messenger ribonucleic acid (mRNA)-1273 vaccine administered into the right arm as an IM injection on Day 1; participants then received Dose 2 of the mRNA-1273 vaccine administered into the right arm as an IM injection at Month 1 and Dose 2 of the 9vHPV vaccine administered into the left arm as an IM injection at Month 6.
- Non-concomitant Group: Participants received Dose 1 of the mRNA-1273 vaccine administered into the right arm as an IM injection on Day 1 and Dose 2 of the mRNA-1273 vaccine administered into the right arm as an IM injection at Month 1. Participants then received Dose 1 of the 9vHPV vaccine administered into the left arm as an IM injection at Month 2 and Dose 2 of the 9vHPV vaccine administered into the left arm as an IM injection at Month 8.
Period: Overall Study
Arm/Group | Concomitant Group | Non-concomitant Group
Started | 82 | 83
Vaccinated: mRNA-1273 Dose 1 | 81 | 81
Vaccinated: 9vHPV Dose 1 | 81 | 72
Vaccinated: mRNA-1273 Dose 2 | 78 | 78
Vaccinated: 9vHPV Dose 2 | 67 | 66
Concomitant Group Dose 1 Day 1: 9vHPV | 81 | 0
Concomitant Group Dose 1 Day 1: mRNA-1273 | 81 | 0
Concomitant Group Dose 2 Month 1: mRNA-1273 | 78 | 0
Concomitant Group Dose 2 Month 6: 9vHPV | 67 | 0
Non-concomitant Group Dose 1 Day 1: mRNA-1273 | 0 | 81
Non-concomitant Group Dose 2 Month 1: mRNA-1273 | 0 | 78
Non-concomitant Group Dose 1 Month 2: 9vHPV | 0 | 72
Non-concomitant Group Dose 2 Month 8: 9vHPV | 0 | 66
Completed | 66 | 64
Not Completed | 16 | 19
Not completed — Randomized by Mistake Without Study Treatment | 0 | 1
Not completed — Withdrawal By Parent/Guardian | 10 | 10
Not completed — Lost to Follow-up | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Group | Non-concomitant Group | Total
Number analyzed (Participants) | 82 | 83 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.9 (0.9) | 9.9 (0.8) | 9.9 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 88
  Male | 39 | 38 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 46 | 96
  Not Hispanic or Latino | 32 | 37 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 31 | 59
  White | 53 | 48 | 101
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of Anti-Human Papillomavirus Vaccine Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 (9vHPV)
Description: Antibodies to HPV types 6/11/16/18/31/33/45/52/58 were measured using a competitive Luminex immunoassay (cLIA). Per protocol, antibody titers were expressed as milli Merck units/milliliter (mMU/mL). Geometric Mean Titers (GMTs) are reported for both arms for all randomized participants included in the per-protocol immunogenicity (PPI) population. The PPI population is HPV-type specific.
Time Frame: Up approximately 4 weeks post vaccination with 9vHPV Dose 2
Population: The analysis population is HPV-type specific; the number of participants analyzed is the total number of participants for inclusion in any HPV type-specific PPI. The type-specific PPI population includes all randomized participants who were seronegative pre 9vHPV vaccination to the relevant HPV type(s); had all protocol planned 9vHPV vaccinations; had evaluable serology results post Dose 2; had no protocol deviations that may affect evaluation of participant's immune response to vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Concomitant Group | Non-concomitant Group
Number analyzed (Participants) | 51 | 49
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 47 | 46
  Anti-HPV 6 | 2198.5 [1806.9 to 2674.8] | 1806.8 [1481.8 to 2202.9]
  Anti-HPV 11: number analyzed (Participants) | 46 | 49
  Anti-HPV 11 | 1517.6 [1247.5 to 1846.2] | 1138.2 [941.4 to 1376.2]
  Anti-HPV 16: number analyzed (Participants) | 47 | 46
  Anti-HPV 16 | 9595.8 [7822.5 to 11771.0] | 7042.3 [5728.2 to 8657.7]
  Anti-HPV 18: number analyzed (Participants) | 48 | 46
  Anti-HPV 18 | 2139.2 [1721.3 to 2658.6] | 1713.2 [1372.1 to 2139.1]
  Anti-HPV 31: number analyzed (Participants) | 46 | 47
  Anti-HPV 31 | 1695.6 [1383.9 to 2077.3] | 1404.7 [1149.0 to 1717.2]
  Anti-HPV 33: number analyzed (Participants) | 48 | 47
  Anti-HPV 33 | 1172.3 [950.8 to 1445.5] | 889.9 [720.2 to 1099.6]
  Anti-HPV 45: number analyzed (Participants) | 50 | 47
  Anti-HPV 45 | 518.0 [413.0 to 649.6] | 370.8 [293.6 to 468.4]
  Anti-HPV 52: number analyzed (Participants) | 49 | 48
  Anti-HPV 52 | 733.6 [614.4 to 875.9] | 504.7 [421.9 to 603.7]
  Anti-HPV 58: number analyzed (Participants) | 48 | 48
  Anti-HPV 58 | 1095.2 [900.5 to 1332.1] | 912.6 [750.3 to 1110.0]
Statistical Analysis 1: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 6; Test type: Other — Geometric Mean Titer (GMT) Ratio with corresponding 2-sided 95% confidence interval (CI) was calculated using an analysis of variance model (ANOVA) with a response of log individual anti-HPV titers and a fixed effect for the vaccination groups, Concomitant Group versus Non-concomitant Group. GMT Ratio is reported for Concomitant Group/Non-concomitant Group; Geometric Mean Titer (GMT) Ratio = 1.22, 95% CI 2-sided [0.92 to 1.61] — GMT Ratio is between Concomitant Group/Non-concomitant Group
Statistical Analysis 2: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 11; Test type: Other — Geometric Mean Titer (GMT) Ratio with corresponding 2-sided 95% confidence interval (CI) was calculated using an analysis of variance model (ANOVA) with a response of log individual anti-HPV titers and a fixed effect for the vaccination groups, Concomitant Group versus Non-Concomitant Group. GMT Ratio is between Concomitant Group/Non-concomitant Group; Geometric Mean Titer (GMT) Ratio = 1.33, 95% CI 2-sided [1.01 to 1.75] — GMT Ratio is between Concomitant Group/Non-concomitant Group
Statistical Analysis 3: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 16; Test type: Other — [test comment as in outcome 1, analysis 2]; Geometric Mean Titer (GMT) Ratio = 1.36, 95% CI 2-sided [1.02 to 1.82] — GMT Ratio is between Concomitant Group/Non-concomitant Group
Statistical Analysis 4: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 18; Test type: Other — Geometric Mean Titer (GMT) Ratio with corresponding 2-sided 95% confidence interval (CI) was calculated using an analysis of variance model (ANOVA) with a response of log individual anti-HPV titers and a fixed effect for the vaccination groups, Concomitant Group versus Non-Concomitant Group. Group. GMT Ratio is between Concomitant Group/Non-concomitant Group; Geometric Mean Titer (GMT) Ratio = 1.25, 95% CI 2-sided [0.92 to 1.70] — GMT Ratio is between Concomitant Group/Non-concomitant Group
Statistical Analysis 5: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 31; Test type: Other — [test comment as in outcome 1, analysis 4]; Geometric Mean Titer (GMT) Ratio = 1.21, 95% CI 2-sided [0.91 to 1.61] — GMT Ratio is between Concomitant Group/Non-concomitant Group
Statistical Analysis 6: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 33; Test type: Other — [test comment as in outcome 1, analysis 2]; Geometric Mean Titer (GMT) Ratio = 1.32, 95% CI 2-sided [0.98 to 1.77] — GMT Ratio is between Concomitant Group/Non-concomitant Group
Statistical Analysis 7: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 45; Test type: Other — [test comment as in outcome 1, analysis 2]; Geometric Mean Titer (GMT) Ratio = 1.40, 95% CI 2-sided [1.01 to 1.93] — GMT Ratio is between Concomitant Group/Non-concomitant Group
Statistical Analysis 8: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 52; Test type: Other — [test comment as in outcome 1, analysis 2]; Geometric Mean Titer (GMT) Ratio = 1.45, 95% CI 2-sided [1.13 to 1.87] — GMT Ratio is between Concomitant Group/Non-concomitant Group
Statistical Analysis 9: Comparison: Concomitant Group vs Non-concomitant Group; Anti-HPV 58; Test type: Other — [test comment as in outcome 1, analysis 2]; Geometric Mean Titer (GMT) Ratio = 1.20, 95% CI 2-sided [0.91 to 1.58] — GMT Ratio is between Concomitant Group/Non-concomitant Group

2. Primary Outcome: Geometric Mean Concentrations of SARS-CoV-2 Spike Protein-Specific Binding Antibodies
Description: The geometric mean concentration (GMC) of serum-derived antibodies to severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) spike protein was determined using an electrochemiluminescence (ECL) assay. GMCs are reported for both arms for all randomized participants included in the mRNA-1273 per-protocol (mRNA-1273-PP) population.
Time Frame: Up approximately 4 weeks post vaccination with mRNA-1273 Dose 2
Population: mRNA-1273-PP population: all randomized participants who; had all protocol planned mRNA-1273 vaccinations; had evaluable serology results post mRNA-1273 Dose 2 vaccination; no protocol deviations that may affect evaluation of participant's immune response to mRNA-1273 vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Concomitant Group | Non-concomitant Group
Number analyzed (Participants) | 56 | 60
μg/mL | 763084.3 [673224.4 to 864938.4] | 650527.9 [576365.9 to 734232.5]
Statistical Analysis 1: Comparison: Concomitant Group vs Non-concomitant Group; Geometric Mean Concentration (GMC) Ratio; Test type: Other — Geometric Mean Concentration (GMC) Ratio with corresponding 2-sided 95% confidence interval (CI) was calculated using an analysis of variance model (ANOVA) with a response of log individual anti-SARS-CoV-2 concentrations and a fixed effect for the vaccination groups, Concomitant Group versus Non-Concomitant Group. GMC Ratio is between Concomitant Group/Non-concomitant Group; Geometric Mean Concentration (GMC) Ratio = 1.17, 95% CI 2-sided [0.99 to 1.40] — GMC Ratio is between Concomitant Group/Non-concomitant Group

3. Primary Outcome: Percentage of Participants With ≥1 Solicited Injection-site Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited AEs are predefined local AEs (at the injection site) for which the participant was specifically questioned, and noted by the participant in their vaccine report card (VRC). Per protocol, the percentage of participants with ≥1 solicited injection site AE has been reported separately based on injection site for participants in the Concomitant Group (Day 1 mRNA-1273 Dose 1 right arm; Day 1 9vHPV Dose 1 left arm; Month 1 mRNA-1273 Dose 2 right arm; Month 6 9vHPV Dose 2 left arm) and Non-Concomitant Group (Day 1 mRNA-1273 Dose 1 right arm; Month 1 mRNA-1273 Dose 2 right arm; Month 2 9vHPV Dose 1 left arm; Month 8 9vHPV Dose 2 left arm). Per protocol, reporting for Concomitant Group Day 1 Dose 1 separated by injection site is specific to this outcome only and does not apply to other safety outcomes.
Time Frame: Up to approximately Day 7 post vaccination with any study vaccine
Population: Per protocol, the safety analyses population consists of all randomized participants who received at least 1 dose of any study vaccine. Participants are included in the treatment group corresponding to the study vaccine they actually received. Per protocol, reporting for Concomitant Group Day 1 Dose 1 separated by injection site is specific to this outcome only and does not apply to other safety outcomes.
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-concomitant Group
Number analyzed (Participants) | 81 | 81
Percentage of Participants
  Concomitant Group: Day 1 -mRNA-1273 Dose 1 (right arm): number analyzed (Participants) | 81 | 0
  Concomitant Group: Day 1 -mRNA-1273 Dose 1 (right arm) | 49.4 |
  Concomitant Group: Day 1 - 9vHPV Dose 1 (left arm): number analyzed (Participants) | 81 | 0
  Concomitant Group: Day 1 - 9vHPV Dose 1 (left arm) | 39.5 |
  Concomitant Group: Month 1 - mRNA-1273 Dose 2 (right arm): number analyzed (Participants) | 78 | 0
  Concomitant Group: Month 1 - mRNA-1273 Dose 2 (right arm) | 35.9 |
  Concomitant Group: Month 6 - 9vHPV Dose 2 (left arm): number analyzed (Participants) | 67 | 0
  Concomitant Group: Month 6 - 9vHPV Dose 2 (left arm) | 26.9 |
  Non-concomitant Group: Day 1 - mRNA-1273 Dose 1 (right arm): number analyzed (Participants) | 0 | 81
  Non-concomitant Group: Day 1 - mRNA-1273 Dose 1 (right arm) |  | 55.6
  Non-concomitant Group: Month 1 -mRNA-1273 Dose 2 (right arm): number analyzed (Participants) | 0 | 78
  Non-concomitant Group: Month 1 -mRNA-1273 Dose 2 (right arm) |  | 44.9
  Non-Concomitant Group: Month 2 - 9vHPV Dose 1 (left arm): number analyzed (Participants) | 0 | 72
  Non-Concomitant Group: Month 2 - 9vHPV Dose 1 (left arm) |  | 29.2
  Non-concomitant Group: Month 8 - 9vHPV Dose 2 (left arm): number analyzed (Participants) | 0 | 66
  Non-concomitant Group: Month 8 - 9vHPV Dose 2 (left arm) |  | 43.9

4. Primary Outcome: Percentage of Participants With ≥1 Solicited Systemic AE
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited AEs are predefined systemic events for which the participant is specifically questioned, and which are noted by the participant in their VRC. Per protocol the percentage of participants who experienced ≥1 solicited systemic (affecting the whole body) AE are reported here for participants in the Concomitant (Day 1 mRNA-1273 Dose 1 right arm + 9vHPV Dose 1 left arm; Month 1 mRNA-1273 Dose 2 right arm; Month 6 9vHPV Dose 2 left arm) and Non-Concomitant Groups (Day 1 mRNA-1273 Dose 1 right arm; Month 1 mRNA-1273 Dose 2 right arm; Month 2 9vHPV Dose 1 left arm; Month 8 9vHPV Dose 2 left arm). Per protocol, reporting is based on time of injection; as 9vHPV Dose 1 AND mRNA-1273 Dose 1 were both given on Day 1 of the Concomitant Group they have been combined below.
Time Frame: Up to approximately Day 7 post vaccination with any study vaccine
Population: Per protocol, the safety analyses population consists of all randomized participants who received at least 1 dose of any study vaccine. Participants are included in the treatment group corresponding to the study vaccine they actually received. Per protocol, reporting is based on time of injection; as 9vHPV Dose 1 AND mRNA-1273 Dose 1 were both given on Day 1 of the Concomitant Group they have been combined below.
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-concomitant Group
Number analyzed (Participants) | 81 | 81
Percentage of Participants
  Concomitant Group: Day 1 - 9vHPV Dose 1 + mRNA-1273 Dose 1: number analyzed (Participants) | 81 | 0
  Concomitant Group: Day 1 - 9vHPV Dose 1 + mRNA-1273 Dose 1 | 33.3 |
  Concomitant Group: Month 1 - mRNA-1273 Dose 2: number analyzed (Participants) | 78 | 0
  Concomitant Group: Month 1 - mRNA-1273 Dose 2 | 33.3 |
  Concomitant Group: Month 6 - 9vHPV Dose 2: number analyzed (Participants) | 67 | 0
  Concomitant Group: Month 6 - 9vHPV Dose 2 | 17.9 |
  Non-concomitant Group: Day 1 - mRNA-1273 Dose 1: number analyzed (Participants) | 0 | 81
  Non-concomitant Group: Day 1 - mRNA-1273 Dose 1 |  | 37.0
  Non-concomitant Group: Month 1 - mRNA-1273 Dose 2: number analyzed (Participants) | 0 | 78
  Non-concomitant Group: Month 1 - mRNA-1273 Dose 2 |  | 33.3
  Non-concomitant Group: Month 2 - 9vHPV Dose 1: number analyzed (Participants) | 0 | 72
  Non-concomitant Group: Month 2 - 9vHPV Dose 1 |  | 16.7
  Non-concomitant Group: Month 8 - 9vHPV Dose 2: number analyzed (Participants) | 0 | 66
  Non-concomitant Group: Month 8 - 9vHPV Dose 2 |  | 10.6

5. Primary Outcome: Percentage of Participants With ≥1 Serious Adverse Event (SAE)
Description: A serious adverse event (SAE) was defined as one that results in death, is life threatening, or requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or other important medical event that may require medical intervention. Per protocol the percentage of participants who experienced ≥1 SAE are reported here for participants in the Concomitant (Day 1 mRNA-1273 Dose 1 right arm + 9vHPV Dose 1 left arm; Month 1 mRNA-1273 Dose 2 right arm; Month 6 9vHPV Dose 2 left arm) and Non-Concomitant Groups (Day 1 mRNA-1273 Dose 1 right arm; Month 1 mRNA-1273 Dose 2 right arm; Month 2 9vHPV Dose 1 left arm; Month 8 9vHPV Dose 2 left arm). Per protocol, reporting is based on time of injection; as 9vHPV Dose 1 AND mRNA-1273 Dose 1 were both given on Day 1 of the Concomitant Group they have been combined below.
Time Frame: Up to approximately Day 28 post vaccination with any study vaccine
Population: Per protocol, the safety analyses population consists of all randomized participants who received at least 1 dose of any study vaccine. Participants are included in thetreatment group corresponding to the study vaccine they actually received. Per protocol, reporting is based on time of injection; as 9vHPV Dose 1 AND mRNA-1273 Dose 1were both given on Day 1 of the Concomitant Group they have been combined below.
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-concomitant Group
Number analyzed (Participants) | 81 | 81
Percentage of Participants
  Concomitant Group: Day 1 - 9vHPV Dose 1 + mRNA-1273 Dose 1: number analyzed (Participants) | 81 | 0
  Concomitant Group: Day 1 - 9vHPV Dose 1 + mRNA-1273 Dose 1 | 0.0 |
  Concomitant Group: Month 1 - mRNA-1273 Dose 2: number analyzed (Participants) | 78 | 0
  Concomitant Group: Month 1 - mRNA-1273 Dose 2 | 0.0 |
  Concomitant Group: Month 6 - 9vHPV Dose 2: number analyzed (Participants) | 67 | 0
  Concomitant Group: Month 6 - 9vHPV Dose 2 | 0.0 |
  Non-concomitant Group: Day 1 - mRNA-1273 Dose 1: number analyzed (Participants) | 0 | 81
  Non-concomitant Group: Day 1 - mRNA-1273 Dose 1 |  | 0.0
  Non-concomitant Group: Month 1 - mRNA-1273 Dose 2: number analyzed (Participants) | 0 | 78
  Non-concomitant Group: Month 1 - mRNA-1273 Dose 2 |  | 0.0
  Non-concomitant Group: Month 2 - 9vHPV Dose 1: number analyzed (Participants) | 0 | 72
  Non-concomitant Group: Month 2 - 9vHPV Dose 1 |  | 0.0
  Non-concomitant Group: Month 8 - 9vHPV Dose 2: number analyzed (Participants) | 0 | 66
  Non-concomitant Group: Month 8 - 9vHPV Dose 2 |  | 0.0

6. Primary Outcome: Percentage of Participants With ≥1 Vaccine-Related SAE
Description: A SAE was defined as one that results in death, is life threatening, or requires hospitalization/prolongation of existing hospitalization, results in persistent/significant disability/incapacity, is a congenital anomaly/birth defect, or other important medical event that may require medical intervention. An SAE judged by the investigator to be related to the study vaccine is a vaccine-related SAE. Per protocol the percentage of participants who experienced ≥1 vaccine-related SAE are reported here for participants in Concomitant (Day 1 mRNA-1273 Dose 1 right arm + 9vHPV Dose 1 left arm; Month 1 mRNA-1273 Dose 2 right arm; Month 6 9vHPV Dose 2 left arm) and Non-Concomitant Groups (Day 1 mRNA-1273 Dose 1 right arm; Month 1 mRNA-1273 Dose 2 right arm; Month 2 9vHPV Dose 1 left arm; Month 8 9vHPV Dose 2 left arm). Per protocol, reporting is based on time of injection; as 9vHPV Dose 1 AND mRNA-1273 Dose 1 were both given on Day 1 of the Concomitant Group they have been combined below.
Time Frame: Up to approximately 9 Months
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-concomitant Group
Number analyzed (Participants) | 81 | 81
Percentage of Participants
  Concomitant Group: Day 1 - 9vHPV Dose 1 + mRNA-1273 Dose 1: number analyzed (Participants) | 81 | 0
  Concomitant Group: Day 1 - 9vHPV Dose 1 + mRNA-1273 Dose 1 | 0.0 |
  Concomitant Group: Month 1 - mRNA-1273 Dose 2: number analyzed (Participants) | 78 | 0
  Concomitant Group: Month 1 - mRNA-1273 Dose 2 | 0.0 |
  Concomitant Group: Month 6 - 9vHPV Dose 2: number analyzed (Participants) | 67 | 0
  Concomitant Group: Month 6 - 9vHPV Dose 2 | 0.0 |
  Non-concomitant Group: Day 1 - mRNA-1273 Dose 1: number analyzed (Participants) | 0 | 81
  Non-concomitant Group: Day 1 - mRNA-1273 Dose 1 |  | 0.0
  Non-concomitant Group: Month 1 - mRNA-1273 Dose 2: number analyzed (Participants) | 0 | 78
  Non-concomitant Group: Month 1 - mRNA-1273 Dose 2 |  | 0.0
  Non-concomitant Group: Month 2 - 9vHPV Dose 1: number analyzed (Participants) | 0 | 72
  Non-concomitant Group: Month 2 - 9vHPV Dose 1 |  | 0.0
  Non-concomitant Group: Month 8 - 9vHPV Dose 2: number analyzed (Participants) | 0 | 66
  Non-concomitant Group: Month 8 - 9vHPV Dose 2 |  | 0.0

7. Secondary Outcome: Percentage of Participants Who Seroconvert to Each of the 9vHPV Vaccine Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 Following Administration of a 2-Dose Regimen of 9vHPV Vaccine
Description: Serum-derived antibodies to HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 were measured with a competitive luminex immunoassay (cLIA). Seroconversion is defined as changing from cLIA anti-HPV seronegative serum antibodies for 9vHPV types at pre-vaccination to cLIA anti-HPV seropositive at 4 weeks post vaccination with 9vHPV Dose 2. A participant with anti-HPV cLIA titer at or above the serostatus cutoff values of the cLIA for a given HPV type is considered seropositive for that HPV type. The serostatus cutoffs (milli Merck units/milliliter (mMU/mL) for HPV types were as follows: HPV Type 6: ≥34, HPV Type 11: ≥25; HPV Type 16: ≥32, HPV Type 18: ≥26, HPV Type 31: ≥15, HPV Type 33: ≥10, HPV Type 45: ≥10, HPV Type 52: ≥14, and HPV Type 58: ≥10. Percentage of participants who seroconverted are reported for both arms for all randomized participants included in the PPI population. The PPI population is HPV-type specific.
Time Frame: Up to approximately 4 weeks post vaccination with 9vHPV Dose 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-concomitant Group
Number analyzed (Participants) | 51 | 49
Percentage of Participants
  Anti-HPV 6 cLIA ≥34 mMU/ mL: number analyzed (Participants) | 47 | 46
  Anti-HPV 6 cLIA ≥34 mMU/ mL | 100.0 [92.5 to 100.0] | 100.0 [92.3 to 100]
  Anti-HPV 11 cLIA ≥25 mMU/ mL: number analyzed (Participants) | 46 | 49
  Anti-HPV 11 cLIA ≥25 mMU/ mL | 100.0 [92.3 to 100.0] | 100.0 [92.7 to 100.0]
  Anti-HPV 16 cLIA ≥32 mMU/ mL: number analyzed (Participants) | 47 | 46
  Anti-HPV 16 cLIA ≥32 mMU/ mL | 100.0 [92.5 to 100.0] | 100.0 [92.3 to 100.0]
  Anti-HPV 18 cLIA ≥26 mMU/ mL: number analyzed (Participants) | 48 | 46
  Anti-HPV 18 cLIA ≥26 mMU/ mL | 100.0 [92.6 to 100.0] | 100.0 [92.3 to 100.0]
  Anti-HPV 31 cLIA ≥15 mMU/ mL: number analyzed (Participants) | 46 | 47
  Anti-HPV 31 cLIA ≥15 mMU/ mL | 100.0 [92.3 to 100.0] | 100.0 [92.5 to 100.0]
  Anti-HPV 33 cLIA ≥10 mMU/ mL: number analyzed (Participants) | 48 | 47
  Anti-HPV 33 cLIA ≥10 mMU/ mL | 100.0 [92.6 to 100.0] | 100.0 [92.5 to 100.0]
  Anti-HPV 45 cLIA ≥10 mMU/ mL: number analyzed (Participants) | 50 | 47
  Anti-HPV 45 cLIA ≥10 mMU/ mL | 100.0 [92.9 to 100.0] | 100.0 [92.5 to 100.0]
  Anti-HPV 52 cLIA ≥14 mMU/ mL: number analyzed (Participants) | 49 | 48
  Anti-HPV 52 cLIA ≥14 mMU/ mL | 100.0 [92.7 to 100.0] | 100.0 [92.6 to 100.0]
  Anti-HPV 58 cLIA ≥10 mMU/ mL: number analyzed (Participants) | 48 | 48
  Anti-HPV 58 cLIA ≥10 mMU/ mL | 100.0 [92.6 to 100.0] | 100.0 [92.6 to 100.0]

8. Secondary Outcome: Percentage of Participants Who Experience Seroresponse Following Administration of a 2-Dose Regimen of mRNA-1273 Vaccine
Description: Serum-derived antibodies to severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) spike protein was determined using an electrochemiluminescence (ECL) assay. Seroresponse is defined as a ≥4-fold rise in SARS-CoV-2 spike protein-specific binding antibody concentration from baseline to 4 weeks post vaccination with mRNA-1273 Dose 2. Percentage of participants who experience seroresponse are reported for both arms for all randomized participants included in the mRNA-1273-PP population.
Time Frame: Up to approximately 4 weeks post vaccination with mRNA-1273 Dose 2
Population: mRNA-1273-PP population: all randomized participants who; received all protocol planned mRNA-1273 vaccinations; had evaluable serology results from samples collected post mRNA-1273 Dose 2 vaccination; no protocol deviations that may affect evaluation of participant's immune response to mRNA-1273 vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-concomitant Group
Number analyzed (Participants) | 56 | 60
Percentage of Participants | 96.4 [87.7 to 99.6] | 95.0 [86.1 to 99.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 9 Months
Description: Population for All-cause mortality was All Randomized Participants. Population for Non-serious adverse events and serious adverse events was All Participants as Treated (APaT). The APaT population consists of all randomized participants who received at least 1 dose of any study vaccine; participants were included in the treatment group corresponding to the study vaccine they actually received.
Arm/Group | Concomitant Group | Non-concomitant Group
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/81
Other Adverse Events (participants affected / at risk) | 55/81 | 59/81
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Group (N=81) | Non-concomitant Group (N=81)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (6) | 20 (25)
Nausea (Gastrointestinal disorders) | 9 (10) | 5 (7)
Chills (General disorders) | 13 (16) | 11 (11)
Fatigue (General disorders) | 23 (32) | 23 (38)
Injection site erythema (General disorders) | 6 (7) | 12 (18)
Injection site pain (General disorders) | 46 (113) | 52 (122)
Injection site swelling (General disorders) | 14 (22) | 18 (27)
Pyrexia (General disorders) | 11 (15) | 10 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 16 (19)
Headache (Nervous system disorders) | 26 (33) | 30 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT05119855/Prot_SAP_000.pdf